CLINICAL TRIAL: NCT05817669
Title: A Phase 2, Randomized, Placebo-controlled, Parallel-group, Double-blinded, proof-of Concept Study to Evaluate the Safety and Efficacy of Intravenous Efgartigimod in Adult Participants With Primary Sjögren's Syndrome
Brief Title: A Study of the Safety and Effectiveness of Efgartigimod in Patients With Primary Sjögren's Syndrome (pSS)
Acronym: rho
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARGX-113-2106; 2021-005911-30 (EudraCT Number)
Record Dates: First submitted 2023-02-01; First posted 2023-04-18 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized to receive efgartigimod 10 mg/kg or placebo in a 2:1 ratio, respectively. All participants will receive efgartigimod IV 10 mg/kg or placebo once weekly for 24 weeks during the treatment period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV arm (Experimental): patients receiving infusions of Efgartigimod IV
  Interventions: Biological: Efgartigimod
- Placebo arm (Placebo Comparator): patients receiving infusions of placebo IV
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Efgartigimod — Patients receiving efgartigimod infusions
  Arms: Efgartigimod IV arm
Biological: Placebo — Patients receiving placebo infusions
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to assess the efficacy and safety of human FcRn blocking therapy with efgartigimod compared to placebo, in participants with pSS.

DETAILED DESCRIPTION:
Primary Sjogren Syndrome (pSS) is an autoimmune disease with still unmet treatment needs. Efgartigimod, a human FcRn antagonist, has the potential to successfully treat pSS and improve disease manifestations by the reduction of IgG autoantibodies and immune complexes in pSS. The study design is randomized, double-blinded, and placebo-controlled to evaluate the effect of efgartigimod administered as an IV infusion compared to placebo. The study consists of a treatment period when all participants will receive infusions of IP/placebo for 24 weeks. At the end of the randomized treatment period, eligible participants may roll over to an OLE study or remain in this study through the end of the 56-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the legal age of consent for clinical trials when signing the informed consent form
* Is capable of providing signed informed consent and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and measures described in the protocol
* Meets the following criteria at screening: ACR/EULAR 2016 pSS who met criteria ≤7 years before screening; ESSDAI ≥5; Anti-Ro/SS-A positive; Residual salivary flow (UWSF rate >0 and/or SWSF rate >0.10)

Exclusion Criteria:

* Known autoimmune disease or any medical condition that, in the investigator's judgment,would interfere with an accurate assessment of clinical symptoms of pSS or puts the participant at undue risk
* History of malignancy unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of IMP.
* Adequately treated participants with the following cancers may be included at any time: Basal cell or squamous cell skin cancer; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological finding of prostate cancer (TNM stage T1a or T1b) Clinically significant uncontrolled active acute or chronic bacterial, viral, or fungal infection
* Positive serum test at screening for an active infection with any of the following: HBV that is indicative of an acute or chronic infection, unless associated with a negative HBsAg or negative HBV DNA test; HCV based on HCV antibody assay unless a negative RNA test is available; HIV based on test results of a CD4 count of <200 cells/mm3 that are associated with an AIDS-defining condition, HIV based on test results of a CD4 count of >200 cells/mm3 not adequately treated with antiviral therapy
* Clinically significant disease, recent major surgery (within 3 months of screening), or intention to have surgery during the study; or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk
* Immunoglobulin G (IgG) levels cannot be below a certain threshold ( 4g/L)
* Positive covid test at study start
* Some of the medications such as vaccines with live components or medicines that may be prescribed cannot be taken either shortly before or during this study
* Current participation in another interventional clinical study or previously participation in an efgartigimod clinical study and treatment with ≥1 dose of IMP
* Known hypersensitivity to IMP or 1 of its excipients
* History (within 12 months of screening) of current alcohol, drug, or medication abuse as assessed by the investigator
* Pregnant or lactating state or intention to become pregnant during the study
* Secondary Sjögren's syndrome overlap syndromes where another confirmed autoimmune rheumatic or systemic inflammatory condition is the primary diagnosis
* Chinese traditional medicine with known immunomodulatory action

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Hungary (2):
  - Debreceni Egyetem, Debrecen
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt., Székesfehérvár
- Universitair Medisch Centrum Groningen , Dept of Rheumatology and Clinical Immunology, Groningen, Netherlands
- Poland (13):
  - Ambulatorium Barbara Bazela, Elblag
  - MCBK Iwona Czajkowska Anna Podrażka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Centrum Medyczne Plejady, Krakow
  - FutureMeds Krakow, Krakow
  - ETG Lublin, Lublin
  - Reumed Spolka z o.o., Lublin
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością Medic-R Sp.k., Poznan
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - MICS Centrum Medyczne Warszawa, Warsaw
  - KO-Med - Centrum Badań Medycznych NIGRiR, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - FutureMeds Targowek, Warsaw
  - FutureMeds Wroclaw, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, double-blinded study was conducted in adult participants with primary Sjögren's disease (pSjD) at 15 investigational sites in 3 countries (Belgium, Hungary, and Poland) between 08-May-2023 and 12-Feb-2024.
Pre-assignment Details: A total of 34 participants were enrolled in the study. The study consisted of screening (≤4 weeks), treatment period (24 weeks), and follow-up period (56 days). Participants were randomized in a 2:1 ratio to either receive efgartigimod or placebo for 24 weeks. At the end of treatment period, eligible participants rolled over to an open-label extension (OLE) study (ARGX-113-2211 [NCT06203457]) or remained in the study for the post-treatment follow-up period.
Groups:
- Efgartigimod: Participants received efgartigimod 10 milligram per kilogram (mg/kg) once weekly via intravenous (IV) infusion for up to 24 weeks.
- Placebo: Participants received placebo matched to efgartigimod once weekly via IV infusion for up to 24 weeks.
Period: Overall Study
Arm/Group | Efgartigimod | Placebo
Started | 23 | 11
Completed (Completed 24-week treatment period) | 20 | 7
Not Completed | 3 | 4
Not completed — Prohibited medication used | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study treatment and who were classified according to the planned treatment.
Groups:
- Efgartigimod: Participants received efgartigimod 10 mg/kg once weekly via IV infusion for up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Efgartigimod | Placebo | Total
Number analyzed (Participants) | 23 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (12.57) | 54.7 (12.42) | 51.6 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 33
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 11 | 33
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Overall CRESS Response of at Least 3 of 5 Items at Week 24
Description: A Composite of Relevant Endpoints for Sjögren's Syndrome (CRESS) responder is defined as improvements in at least 3 of the 5 items of CRESS (systemic disease activity, patient-reported symptoms, tear gland function, salivary gland function and serology. The score ranges from 0 to 9 (higher score = worse symptoms).
Time Frame: Week 24
Population: The Efficacy Analysis Set (EAS) included all participants eligible for efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 45.5 [26.92 to 65.34] | 11.1 [1.99 to 43.50]

2. Secondary Outcome: Number of Participants With TEAEs, AESI, and SAEs
Description: A treatment-emergent adverse event (TEAE): adverse events reported from the first dose up to and including 60 days after the final dose were considered treatment-emergent. Serious adverse event (SAE): adverse event that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or other situations. Adverse event of special interest (AESI): adverse event related to 'Infections and infestations'.
Time Frame: Up to 32 weeks
Population: The Safety Analysis Set (SAF) included all participants exposed to the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Any TEAE | 20 | 7
  Any AESI | 15 | 5
  Any SAE | 1 | 0

3. Secondary Outcome: Percentage of Participants With MCII in ESSDAI at Week 24
Description: European Alliance of Associations for Rheumatology (EULAR) Sjögren's Syndrome Disease Activity Index (ESSDAI) measures systemic disease activity in participants with pSjD and consists of 11 organ-specific domains and 1 biological domain that contribute to disease activity level scoring. Each domain is given a certain weight, which gives a score between 0 and 123 (higher score =worse symptoms). Minimally clinically important improvement (MCII) in ESSDAI was defined as improvement of at least 3 points in ESSDAI score at Week 24.
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 72.7 [51.85 to 86.85] | 55.6 [26.67 to 81.12]

4. Secondary Outcome: Percentage of Participants With Low Disease Activity in ESSDAI at Week 24
Description: ESSDAI measures systemic disease activity in participants with pSjD and consists of 11 organ-specific domains and 1 biological domain that contribute to disease activity level scoring. Each domain is given a certain weight, which gives a score between 0 and 123 (higher score =worse symptoms). Low disease activity in ESSDAI was defined as ESSDAI score of less than 5 at Week 24.
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 59.1 [38.73 to 76.74] | 22.2 [6.32 to 54.74]

5. Secondary Outcome: Percentage of Participants With MCII in clinESSDAI at Week 24
Description: Clinical (clin)ESSDAI includes the same 11 organ-specific domains as ESSDAI but with different domain weighting and without the biological domain. This way any change in clinESSDAI score would reflect disease specific features, irrespective of B-cell activity. The clinESSDAI score ranges between 0-135 (higher score = worse symptoms). Minimal clinically important improvement (MCII) in clinESSDAI was defined as improvement of at least 3 points in clinESSDAI score at Week 24.
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 77.3 [56.56 to 89.88] | 77.8 [45.26 to 93.68]

6. Secondary Outcome: Percentage of Participants With Low Disease Activity in clinESSDAI at Week 24
Description: clinESSDAI includes the same 11 organ-specific domains as ESSDAI but with different domain weighting and without the biological domain. This way any change in clinESSDAI score would reflect disease specific features, irrespective of B-cell activity. The clinESSDAI score ranges between 0-135 (higher score = worse symptoms). Low disease activity in clinESSDAI was defined as clinESSDAI score of less than 5 at Week 24.
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 59.1 [38.73 to 76.74] | 33.3 [12.06 to 64.58]

7. Secondary Outcome: Percentage of Participants With MCII in ESSPRI at Week 24
Description: Minimal clinically important improvement in ESSPRI was defined as decrease of 1 point or at least ≥15% at Week 24. ESSPRI is a questionnaire that has been developed to measure self-reported symptoms in participants with pSjD. The score ranges from 0 (no symptoms) to 10 (more symptoms).
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 31.8 [16.36 to 52.68] | 33.3 [12.06 to 64.58]

8. Secondary Outcome: Change From Baseline in ESSDAI Score at Week 24
Description: ESSDAI measures systemic disease activity in participants with pSjD and consists of 11 organ-specific domains and 1 biological domain that contribute to disease activity level scoring. Each domain is given a certain weight, which gives a score between 0 and 123 (higher score = worse symptoms).
Time Frame: Baseline (Day 1) and Week 24
Population: EAS - Only participants with data collected at baseline and Week 24 are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 19 | 7
score on a scale | -5.0 [-10.0 to -4.0] | -4.0 [-13.0 to -1.0]

9. Secondary Outcome: Change From Baseline in clinESSDAI Score at Week 24
Description: clinESSDAI includes the same 11 organ-specific domains as ESSDAI but with different domain weighting and without the biological domain. This way any change in clinESSDAI score would reflect disease specific features, irrespective of B-cell activity. The clinESSDAI score ranges between 0-135 (higher score = worse symptoms).
Time Frame: Baseline (Day 1) and Week 24
Population: EAS - Only participants with data collected at baseline and Week 24 are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 19 | 7
score on a scale | -7.0 [-12.0 to -3.0] | -4.0 [-17.0 to -3.0]

10. Secondary Outcome: Change From Baseline in ESSPRI Score at Week 24
Description: ESSPRI is a questionnaire that has been developed to measure self-reported symptoms in participants with pSjD. The score ranges from 0 (no symptoms) to 10 (more symptoms).
Time Frame: Baseline (Day 1) and Week 24
Population: EAS - Only participants with data collected at Baseline and Week 24 are reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 16 | 6
score on a scale | -0.500 [-1.333 to 0.333] | -0.833 [-1.333 to -0.333]

11. Secondary Outcome: Percentage of Participants With STAR Score of at Least 5 at Week 24
Description: Sjögren's Tool for Assessing Response (STAR) is a composite endpoint assessing multiple clinically relevant disease features. A STAR responder is defined as a score of at least 5 points. Due to the weighting, participants must be a responder on either systemic disease activity (ESSDAI), patient-reported symptoms (ESSPRI), or both to be an overall STAR responder. The score ranges between 0 and 9 (higher score = worse outcome).
Time Frame: Week 24
Population: EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 22 | 9
Percentage of participants | 54.5 [34.66 to 73.08] | 33.3 [12.06 to 64.58]

12. Secondary Outcome: Plasma Concentration of Efgartigimod
Description: Serum samples were collected at indicated time points to assess the pharmacokinetic (PK) profile of efgartigimod.
Time Frame: Pre-dose at Day 1, Weeks 1, 2, 4, 8, 12, 16, and 20; 30 minutes post-dose at Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: PK population included all randomized participants who received at least 1 dose of efgartigimod and had at least 1 measured concentration of efgartigimod at a scheduled PK time point. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Efgartigimod
Number analyzed (Participants) | 23
Nanograms per milliliter (ng/mL)
  Day 1: Pre-dose | NA (NA) — Mean and standard deviation could not be calculated as the values were below the lower limit of quantification (LLOQ). LLOQ was 200 ng/mL.
  Day 1: 30 minutes post-dose | 179391 (79751)
  Week 1: Pre-dose: number analyzed (Participants) | 22
  Week 1: Pre-dose | 17238 (37356)
  Week 1: 30 minutes post-dose | 187300 (73091)
  Week 2: Pre-dose: number analyzed (Participants) | 22
  Week 2: Pre-dose | 22470 (42838)
  Week 2: 30 minutes post-dose: number analyzed (Participants) | 21
  Week 2: 30 minutes post-dose | 205148 (52448)
  Week 4: Pre-dose: number analyzed (Participants) | 16
  Week 4: Pre-dose | 38595 (65900)
  Week 4: 30 minutes post-dose: number analyzed (Participants) | 16
  Week 4: 30 minutes post-dose | 206414 (102089)
  Week 8: Pre-dose: number analyzed (Participants) | 19
  Week 8: Pre-dose | 14193 (5753)
  Week 8: 30 minutes post-dose: number analyzed (Participants) | 19
  Week 8: 30 minutes post-dose | 203505 (89762)
  Week 12: Pre-dose: number analyzed (Participants) | 18
  Week 12: Pre-dose | 13096 (4523)
  Week 12: 30 minutes post-dose: number analyzed (Participants) | 18
  Week 12: 30 minutes post-dose | 200856 (138766)
  Week 16: Pre-dose: number analyzed (Participants) | 19
  Week 16: Pre-dose | 12676 (5835)
  Week 16: 30 minutes post-dose: number analyzed (Participants) | 19
  Week 16: 30 minutes post-dose | 261647 (215940)
  Week 20: Pre-dose: number analyzed (Participants) | 16
  Week 20: Pre-dose | 12942 (4472)
  Week 20: 30 minutes post-dose: number analyzed (Participants) | 16
  Week 20: 30 minutes post-dose | 194944 (81722)
  Week 24: 30 minutes post-dose: number analyzed (Participants) | 15
  Week 24: 30 minutes post-dose | 14284 (4987)

13. Secondary Outcome: Percentage Change From Baseline in Total IgG Levels in Serum at Week 24
Description: Blood samples were collected at indicated timepoints to assess the total Immunoglobulin (Ig)G levels in serum.
Time Frame: Baseline (Day 1) and Week 24
Population: SAF - Only participants with data available at baseline and Week 24 are reported.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 20 | 7
Percentage change | -57.172 (17.7376) | 0.279 (9.5193)

14. Secondary Outcome: Number of Participants With ADA Against Efgartigimod in Serum
Description: Blood samples were collected to assess anti-drug antibodies (ADAs) against efgartigimod. Treatment-boosted ADA was defined as participants who had a baseline positive sample and the titer value increased 4-fold or more compared to baseline. Treatment-induced ADA was defined as participants who had a baseline negative sample and at least 1 positive post-baseline samples. Treatment-unaffected ADA was defined as participants who had a baseline positive sample, but the titer value did not increase 4-fold or more compared to baseline.
Time Frame: Up to Week 24
Population: SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod | Placebo
Number analyzed (Participants) | 23 | 11
Participants
  Treatment-boosted ADA | 1 | 0
  Treatment-induced ADA | 2 | 0
  Treatment-unaffected ADA | 11 | 3

ADVERSE EVENTS:
Time Frame: Up to 32 weeks.
Description: The SAF included all participants exposed to the study treatment. Any abnormal laboratory results or changes in vital signs are captured in the adverse event listings.
Arm/Group | Efgartigimod | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/11
Other Adverse Events (participants affected / at risk) | 20/23 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=23) | Placebo (N=11)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efgartigimod (N=23) | Placebo (N=11)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT05817669/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT05817669/SAP_001.pdf